CLINICAL TRIAL: NCT02733211
Title: An Open-label, Two-center, Randomized, Cross-over Study to Evaluate the Safety and Efficacy of Night Closed-loop Control Using the MD-Logic Automated Insulin Delivery System Compared to Sensor Augmented Pump Therapy in Poorly Controlled Patients With Type 1 Diabetes at Home
Brief Title: Cross-over Study to Evaluate the Safety and Efficacy of Night Closed-loop Control Using the MD-Logic Automated Insulin Delivery System Compared to Sensor Augmented Pump Therapy in Poorly Controlled Patients With Type 1 Diabetes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Finally it was decided not to initiate the study due to logistical issues
Sponsor: Rabin Medical Center (Other)
Collaborators: GIF (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RMC010016Ctil
Record Dates: First submitted 2016-04-05; First posted 2016-04-11 (Estimated); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Type 1 Diabetes
Keywords: Closed Loop
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Closed Loop System (Experimental): MD-Logic automated insulin delivery system - all subjects wearing the study system during nights over 4 weeks
  Interventions: Device: MD- Logic Closed Loop System
- Sensor augmented pump therapy (Active Comparator): Sensor augmented pump therapy - all subjects are using sensor augmented pump therapy over 4 weeks
  Interventions: Device: sensor augmented pump therapy

INTERVENTIONS:
Device: MD- Logic Closed Loop System — Closed Loop System
  Arms: Closed Loop System
Device: sensor augmented pump therapy — Sensor augmented pump therapy
  Arms: Sensor augmented pump therapy

SUMMARY:
The MD-Logic Automated Insulin Delivery System is intended for patients with type 1 diabetes mellitus for subcutaneous infusion of insulin and the continuous measurement of interstitial glucose to aid in the management of their diabetes. The product automatically adjusts basal insulin delivery and delivers correction boluses in response to real-time glucose measurements by CGM to maintain blood glucose within the desired range, to improve metabolic control without increasing the risk of hypoglycemia.

The proposed study is an open-label, two-center, randomized, cross-over study to evaluate the safety and efficacy of night closed-loop control using the MD-Logic automated insulin delivery system compared to sensor augmented pump therapy in poorly controlled patients with type 1 diabetes at home The objective of this pilot study is to evaluate the safety and efficacy of 4 weeks glucose control using the MD-Logic System in individuals with poorly controlled type 1 diabetes at patient's home

ELIGIBILITY:
Inclusion Criteria:

* Subject with type 1 diabetes >1year since diagnosis
* Insulin infusion pump (CSII) therapy for at least 3 months
* Patients able to use sensor after training based on researcher's estimation
* Age between 10 and 18 years (both included)
* HbA1c at inclusion between 7.5 and 11.0 % (both included)
* Patients willing to follow study instructions
* Patients live with at least one other adult person
* Body Mass Index Standard Deviation Score - below the 95th percentile for age
* Patients with caregivers who are capable of operating a computer based system

Exclusion Criteria:

* Concomitant diseases that influence metabolic control (e.g. anemia, significantly impaired hepatic function, renal failure, history of adrenal insufficiency) or other medical condition, which in the Investigator's opinion, may compromise patient safety Participation in any other interventional study
* Known or suspected allergy to trial products such as adhesives, tapes, needles. An allergy to contrast medium, use of other active medical devices and planned imaging
* Any significant diseases or conditions including psychiatric disorders and substance abuse that, in the opinion of the investigator, is likely to affect the subject's ability to complete the study, or compromise patient safety
* Diabetic ketoacidosis in the past 1 month
* Severe hypoglycemia six month prior to enrollment
* Current use of the following medications: medications that are used to lower blood glucose , Beta blockers, glucocorticoids and other medications, which in the judgment of the investigator would be a contraindication to participation in the study
* Subject is participating in another drug or device study that could affect glucose measurements or glucose management
* Female subject who is pregnant or breast-feeding or is planning to become pregnant within the planned study duration
* Not sufficient vision or hearing to recognize pump/sensor alarms or to perform Blood Glucose-self measurements 4-times daily.
* Relevant severe organ disorders (diabetic nephropathy, diabetic retinopathy, diabetic foot syndrome) or any secondary disease or complication of diabetes mellitus -Subject has unstable or rapidly progressive renal disease or is receiving dialysis-
* Subject has active proliferating retinopathy
* Active gastroparesis
* Patient suffers from an eating disorder

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2019-03 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of glucose sensor readings within 70 to 180 mg/dl (3.9 to 10 mmol/l) during the night (23:00-7:00 h) | At the final visit- Day 115

SECONDARY OUTCOMES:
Percentage of glucose sensor readings within 70 to 180 mg/dl (3.9 to 10 mmol/l) per 24 hours | At the final visit- Day 115
Percentage of glucose sensor readings below 70 mg/dl (3.9 mmol/l) during the night (23:00-7:00 h) and per 24 hours | At the final visit- Day 115
Percentage of glucose sensor readings above 180 mg/dl (10 mmol/l) during the night (23:00-7:00 h) and per 24 hours | At the final visit- Day 115
Average and standard deviation of glucose sensor readings per 24 hours | At the final visit- Day 115
Fasting blood glucose levels | At the final visit- Day 115
HbA1c change from baseline to the end of the intervention period | At the final visit- Day 115
Acceptance and use intention of an Artificial Pancreas | At the final visit- Day 115
  Questionnaire assessing the acceptance and use intention of an Artificial Pancreas
Well-Being | At the final visit- Day 115
  Questionnaire assessing the well-being of participants
Diabetes-specific family conflicts | At the final visit- Day 115
  Questionnaire assessing the diabetes-specific family conflicts of participants
Area under the curve of glucose readings <50 | At the final visit- Day 115
Area under the curve of glucose readings <70 | At the final visit- Day 115
Area under the curve of glucose readings <60 | At the final visit- Day 115
Percentage of glucose readings <70 mg/dl | At the final visit- Day 115
Percentage of glucose readings <60 mg/dl | At the final visit- Day 115
Number of sensor based hypoglycemic events <70mg/dl | At the final visit- Day 115
Number of sensor based hypoglycemic events <60mg/d | At the final visit- Day 115
Number of sensor based hypoglycemic events <50mg/d | At the final visit- Day 115
Area Under the Curve of sensor glucose readings >240 mg/dl | At the final visit- Day 115
Area Under the Curve of sensor glucose readings >300 mg/dl | At the final visit- Day 115
Percentage of sensor glucose readings >240 mg/dl | At the final visit- Day 115
Percentage of sensor glucose readings >300 mg/dl | At the final visit- Day 115

CONTACTS AND LOCATIONS:
Locations (2):
- Diabetes -Zentrum fuer kinder und jugendliche, Hanover, Germany
- Schneider Children's Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No